CLINICAL TRIAL: NCT02894294
Title: Measuring the Impact of Seasonal Malaria Chemoprevention as Part of Routine Malaria Control in Kita, Mali
Brief Title: Evaluation of Seasonal Malaria Chemoprevention in Kita
Status: Completed | Type: Observational
Sponsor: University of Bamako (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alassane Dicko, Professor, University of Bamako
Other Study IDs: FMPOS 2014-70
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Malaria; Anemia
Keywords: malaria; chemoprevention; season; anemia; impact; coverage; children
MeSH Terms: conditions — Malaria; Anemia; Tooth, Impacted

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention district: implementation of the seasonal malaria chemoprevention
  Interventions: Other: implementation of seasonal malaria chemoprevention
- Control district: no implementation of the seasonal malaria chemoprevention

INTERVENTIONS:
Other: implementation of seasonal malaria chemoprevention — administration of therapeutic doses of antimalarials (Sulfadoxine-pyrimethamine [SP] + Amodiaquine [AQ]) at monthly intervals during the high malaria transmission season in children 3-59 months of age.
  Groups: Intervention district

SUMMARY:
Seasonal malaria chemoprevention (SMC) is a new strategy recommended by World Health Organization in 2012 for areas of highly seasonal transmission such as the Sahel. Although randomized controlled trials have shown SMC to be highly effective, evidence and experience from routine implementation of SMC has been lacking. For these reasons, we conducted a comprehensive evaluation of the coverage, adherence, and impact of SMC on malaria infection and disease and anemia when delivered through routine programs using existing community health workers in the Kayes region in Mali. Our evaluation used a pre-post design with cross-sectional surveys and abstraction of routine health information system data in an intervention district (Kita) where SMC was implemented through the health system, and a comparison district (Bafoulabe) where SMC was not implemented.

DETAILED DESCRIPTION:
Seasonal malaria chemoprevention (SMC) is a new strategy recommended by World Health Organization in 2012 for areas of highly seasonal transmission such as the Sahel. Although randomized controlled trials (RCTs) have shown SMC to be highly effective, evidence and experience from routine implementation of SMC has been lacking. For these reasons, we conducted a comprehensive evaluation of the coverage, adherence, and impact of SMC on malaria infection and disease, and anemia when delivered through routine programs using existing community health workers in the Kayes region in Mali. A pre-post design was used, with one intervention district, Kita where four rounds of SMC with Sulfadoxine-Pyrimethamine plus Amodiaquine (SP+AQ) took place in August-November 2014, and one comparison district, Bafoulabe. Cross-sectional surveys were carried out in children aged 3-59 months from 30 randomly selected localities (15/district) at baseline and in follow-up to assess the impact of SMC on malaria parasitemia, fever, malaria illness, and anemia. The baseline survey was performed in July 2014 prior to the start of SMC implementation and the post-intervention (follow-up) surveys took place in December 2014. Blood samples were collected for thick/thin smears for malaria and hemoglobin measurement in two cross-sectional surveys, one prior to SMC in July 2014 and one after SMC in December 2014. The impact on malaria morbidity was assessed using routine data on confirmed malaria cases extracted from the registers by the research team in nine of the 47 community health centers in Kita and seven of the 24 health centers in Bafoulabe. Cross-sectional surveys were also carried out about 7 days after each of the four rounds of SMC to assess caregivers' adherence to the administration of SMC drugs and determine the frequency of adverse events in the intervention district of Kita. Coverage was assessed by cross-sectional in children 3-59 months in 30 randomly selected clusters in the district of Kita using interview of the caregivers and information on the SMC card in December 2014.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3-59 months
* Residence in the study areas
* Provision of inform consent

Exclusion Criteria:

* Age < 3 months or >= 60 months
* Not resident in the study areas
* No provision of inform consent

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-59 months of age
Sampling Method: Probability Sample
Enrollment: 1162 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Coverage of SMC | Four months (August to November in 2014)
  Proportion of the children aged 3-59 months at the time of SMC who received the three days' treatment of SMC during that specific round
Change in malaria infection from baseline | December 2014 (one month post last round of SMC)
  Malaria infection was defined as presence of malaria parasitemia by blood smear
Change in prevalence of malaria illness from baseline | December 2014 (one month post last round of SMC)
  axillary temperature >= 37.5o C and blood smear positive for asexual forms of malaria parasites
Adherence to SMC | 1-3 days post post first SMC dose
  proportion of children who received the second and third dose of AQ at home

SECONDARY OUTCOMES:
Confirmed malaria cases | six months (July to December)
  clinical malaria cases confirmed by rapid diagnostic test or blood smear in the selected health facilities
Change in prevalence of anemia at baseline | December 2014 (one month post last round of SMC)
  hemoglobin < 8 g/dL
Adverse events | 7 days post SMC round in August, September, October and November in 2014
  frequency of adverse events
Change from baseline in frequency of molecular markers of resistance to SP and AQ | December 2014 (one month post last round of SMC)
  mutations at codons 51, 59, and 108 of the dhfr gene, 437 and 540 of the dhps gene, mutations at codon 76 in the P. falciparum chloroquine transporter gene (pfcrt), and at codon 86 of the P. falciparum multidrug resistance gene one (pfmdr1)

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request to the Principal Investigator

REFERENCES:
- [Derived] Diawara F, Steinhardt LC, Mahamar A, Traore T, Kone DT, Diawara H, Kamate B, Kone D, Diallo M, Sadou A, Mihigo J, Sagara I, Djimde AA, Eckert E, Dicko A. Measuring the impact of seasonal malaria chemoprevention as part of routine malaria control in Kita, Mali. Malar J. 2017 Aug 10;16(1):325. doi: 10.1186/s12936-017-1974-x. PMID 28797263